CLINICAL TRIAL: NCT06594133
Title: Longitudinal and Cross-sectional Analysis of Pulmonary Microbiota in Lung Transplant Recipients Infected With Nocardia: A Single-center Retrospective Study
Brief Title: Longitudinal and Cross-sectional Analysis of Pulmonary Microbiota in Lung Transplant Recipients Infected With Nocardia
Acronym: NocardiaLM
Status: Completed | Type: Observational
Sponsor: Zhibin Xu (Other)
Responsible Party: Sponsor-Investigator, Zhibin Xu, Professor of Microbiology, Guangzhou Institute of Respiratory Disease
Organization: Guangzhou Institute of Respiratory Disease (Other)
Other Study IDs: ES-2024-K144
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Nocardia Infections; Lung Transplantation
Keywords: Nocardia;; Pulmonary Microbiota;; Retrospective Study;; Immunosuppression
MeSH Terms: conditions — Nocardia Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Bronchoalveolar lavage fluid (BALF) and blood samples collected from lung transplant recipients. These samples will be used for microbial community analysis and to assess the impact of Nocardia infection on pulmonary and systemic microbiota.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Nocardia Pneumonia Group (NPG): This group consists of lung transplant recipients diagnosed with Nocardia pneumonia. The patients in this group are studied to assess the impact of Nocardia infection on the pulmonary microbiota. Samples including bronchoalveolar lavage fluid (BALF) and blood are collected for microbial community analysis.
  Interventions: Drug: Antibiotic Treatment
- Non-Nocardia Infection Group (NNIG): This group consists of lung transplant recipients who are not infected with Nocardia. These patients serve as the control group and are matched with the Nocardia pneumonia group based on clinical characteristics such as age, sex, and underlying conditions.

INTERVENTIONS:
Drug: Antibiotic Treatment — For lung transplant recipients with Nocardia infection, the treatment regimen could include:
  Sulfamethoxazole/Trimethoprim (Bactrim): 800 mg/160 mg orally or intravenously twice daily for at least 6 months.
  Imipenem: 500 mg intravenously every 6 hours for severe cases. Monitoring: Regular monitoring of blood levels of the drug to avoid toxicity and adjust doses accordingly.
  Groups: Nocardia Pneumonia Group (NPG)

SUMMARY:
This retrospective observational study aims to explore the impact of Nocardia infection on the pulmonary microbiota of lung transplant recipients (LTRs). The study will analyze both cross-sectional and longitudinal data from patients diagnosed with Nocardia pneumonia, comparing microbial composition and diversity between infected and non-infected groups. This research seeks to provide insights into the relationship between pulmonary microbiota alterations and clinical outcomes in LTRs.

DETAILED DESCRIPTION:
This study is a single-center, retrospective, observational study designed to investigate the impact of Nocardia infection on the pulmonary microbiota of lung transplant recipients (LTRs). The study will include both cross-sectional and longitudinal analyses. In the cross-sectional study, 17 LTRs diagnosed with Nocardia pneumonia (Nocardia pneumonia group, NPG) will be compared with 51 non-infected LTRs (non-Nocardia infection group, NNIG) matched for age, sex, and underlying conditions.

The longitudinal study will follow LTRs over a 4-month period, collecting samples before, during, and after treatment. Patients in this group will be categorized into the Recovered group (RG) or Not Recovered group (NRG) based on treatment outcomes. The study will also include a subgroup analysis of patients with disseminated Nocardia infection, comparing pulmonary and systemic microbiota changes.

Microbial diversity and composition will be assessed using high-throughput sequencing of bronchoalveolar lavage fluid (BALF) samples. Statistical analyses will include the Kolmogorov-Smirnov test, ANOVA, and Kruskal-Wallis test for group comparisons, with linear mixed-effects models used to analyze changes over time.

The goal of this study is to provide a deeper understanding of how Nocardia infection affects the pulmonary microbiota in LTRs and to identify key microbial species associated with clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Lung transplant recipients
* Diagnosed with Nocardia pneumonia (for the study group)
* Age ≥ 18 years

Exclusion Criteria:

* Patients with incomplete medical records
* Patients who survived ≤ 3 days after transplantation
* Patients lost to follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study includes lung transplant recipients treated at Guangzhou Medical University First Affiliated Hospital from January 2023 to August 2024, including patients diagnosed with Nocardia pneumonia and matched non-infected controls.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Pulmonary Microbiota Diversity in Nocardia-infected Lung Transplant Recipients | January 2023 to August 2024
  Measurement of alpha and beta diversity of the pulmonary microbiota in BALF samples from lung transplant recipients with and without Nocardia infection. Alpha diversity will be quantified using Shannon diversity index and observed species richness, while beta diversity will be analyzed using Bray-Curtis dissimilarity. Microbial composition and relative abundance will be compared between the Nocardia pneumonia group and the non-Nocardia infection group. Changes in diversity metrics will be analyzed over time to assess the impact of Nocardia infection on pulmonary microbiota.

SECONDARY OUTCOMES:
Correlation Between Pulmonary Microbiota and Clinical Outcomes | January 2023 to August 2024
  Correlation between pulmonary microbiota diversity and clinical factors such as age, kidney function, nutritional status, and immunosuppressive therapy in lung transplant recipients. The analysis includes changes in pulmonary microbiota before and after treatment in patients with Nocardia infection and the number of participants showing significant correlations between microbiota diversity and clinical outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou Institute of Respiratory Diseases, the First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hemmersbach-Miller M, Catania J, Saullo JL. Updates on Nocardia Skin and Soft Tissue Infections in Solid Organ Transplantation. Curr Infect Dis Rep. 2019 Jun 21;21(8):27. doi: 10.1007/s11908-019-0684-7. PMID 31227922
- [Result] Fatahi-Bafghi M. Nocardiosis from 1888 to 2017. Microb Pathog. 2018 Jan;114:369-384. doi: 10.1016/j.micpath.2017.11.012. Epub 2017 Nov 13. PMID 29146497
- [Result] Restrepo A, Clark NM; Infectious Diseases Community of Practice of the American Society of Transplantation. Nocardia infections in solid organ transplantation: Guidelines from the Infectious Diseases Community of Practice of the American Society of Transplantation. Clin Transplant. 2019 Sep;33(9):e13509. doi: 10.1111/ctr.13509. Epub 2019 Mar 19. PMID 30817024
- [Result] Lebeaux D, Morelon E, Suarez F, Lanternier F, Scemla A, Frange P, Mainardi JL, Lecuit M, Lortholary O. Nocardiosis in transplant recipients. Eur J Clin Microbiol Infect Dis. 2014 May;33(5):689-702. doi: 10.1007/s10096-013-2015-5. Epub 2013 Nov 23. PMID 24272063
- [Result] Peleg AY, Husain S, Qureshi ZA, Silveira FP, Sarumi M, Shutt KA, Kwak EJ, Paterson DL. Risk factors, clinical characteristics, and outcome of Nocardia infection in organ transplant recipients: a matched case-control study. Clin Infect Dis. 2007 May 15;44(10):1307-14. doi: 10.1086/514340. Epub 2007 Apr 3. PMID 17443467